CLINICAL TRIAL: NCT02134145
Title: Usability Study of the Scanadu Scout
Brief Title: Scanadu Consumer Health Outcomes (SCOUT) Study
Acronym: SCOUT
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Scanadu, Inc. (Industry)
Responsible Party: Principal Investigator, Steven Steinhubl, Director, Digital Medicine, Scripps Translational Science Institute
Other Study IDs: Scanadu
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Disorder Characterized by Fever
Keywords: Mobile Health; mHealth; Technology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Self Selected Investors: A self selected crowdfunding backers from teh Scanadu Scout Crowdfunding campaign.

SUMMARY:
There is a great need within healthcare to develop systems of care that better engage and activate people in their own care before they become patients. By so doing lay users will be empowered to take charge of their own care in recognizing they can change their health and improve their quality of life. Mobile health technologies such as the Scanadu ScoutTM hold the potential to truly engage individuals in the way needed through real-time data capture, transmission and connectivity.

We propose to evaluate the real-world use of the Scanadu ScoutTM by a cohort of self-selected investors in an earlier crowdfunding campaign on Indiegogo for the Scanadu Scout™, through a prospective observational study. Using validated survey tools and through the remote tracking of frequency of use and physiological measurements from the Scanadu Scout™ device and app.

Participants will receive web-based surveys at 4 time points: baseline, 3, 12 and 18 months.

Participants will be instructed to use the Scanadu Scout™ as much as they would like. The parameters that will be functional on the device and available for measurement by the participant are:

* Heart rate
* Respiratory rate
* Temperature
* Oxygen saturation
* Heart rate variability
* Blood pressure

Data analysis will examine individual participant and aggregate level:

1. Usage and physiologic measurement data of the device,
2. Perceptions of the device, and
3. Changes in self-reported health self-management, health-related quality of life, participant- physician communication and medication adherence between baseline and follow-up.

DETAILED DESCRIPTION:
We propose to evaluate the real-world use of the Scanadu ScoutTM by a cohort of self-selected investors in an earlier crowdfunding campaign on Indiegogo for the Scanadu Scout™, through a prospective observational study. Using validated survey tools and through the remote tracking of frequency of use and physiological measurements from the Scanadu Scout™ device and app, this study will provide preliminary evidence for:

1. Level of engagement and impact of Scanadu ScoutTM on health behavior with a focus on potential risks and safety.
2. Long term (up to 18 months) recurrent usage rate of the various physiologic measurements linked to users and survey data.
3. Ease of use and acceptance of the Scanadu ScoutTM technology.

This study will utilize a longitudinal cohort design. All Scanadu Scout investors (~5000 individuals) will be invited to participate in the study prior to receiving their Scanadu Scout™. Potential participants will receive a link to an online study platform. The platform will contain the Informed Consent form and all the study materials. After a participant reads and signs the Consent the participant will be enrolled in the study and a Scanadu Scout™ device will be sent. The participant will download the Scanadu Scout™ app from the App Stores (iOS/Android). The app will require a handshake with a Scanadu Scout™ device before it becomes fully functional to limit access to study participants.

After signing the Informed Consent form the participant will be asked to complete baseline surveys to assess participant characteristics, health self-management and health-related quality of life prior to using the Scanadu Scout™. At 3 months, 12 months, and at 18 months, a participant will be asked to complete Health Self-Management and Health-Related QOL surveys as well as an additional assessment of their perceptions of the device. Backers who do not wish to partake in this study will not receive the device and will be entitled to get their contribution back.

Participants will be instructed to use the device as much as they would like over the course of the study. The parameters that will be functional on the device and available for measurement by the participant are:

* Heart rate
* Respiratory rate
* Temperature
* Oxygen saturation
* Heart rate variability
* Blood pressure

Data analysis will examine individual participant and aggregate level:

1. Usage and physiologic measurement data of the device,
2. Perceptions of the device, and
3. Changes in self-reported health self-management, health-related quality of life, participant- physician communication and medication adherence between baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Signed Informed Consent Form

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a select cohort of crowdfunding backers for the Scanadu Scout Crowdfunding campaign.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Participant Characteristics | Baseline
  1. Device usage and specific parameter usage
  2. Use of new technology
Changes in psychological outcomes as measured by: | Baseline, 3 months, 12 months, and 18 months
  a. Anxiety Levels (Speilberger State-Trait Anxiety Inventory; STAI Y-6 item)
Changes in Health Outcomes as measured by: | Baseline, 3 months, 12 months, and 18 months
  1. Patient Activation
  2. Health-Related Quality of Life
Changes in Lifestyle Outcomes as measured by: | 3 months, 12 months, and 18 months
  1. Medications
  2. Food Screener
  3. Exercise
  4. Health Communication
Perceptions of the Scanadu Scout™ as measured by | 3 months, 12 months, and 18 months
  1. Satisfaction with technology (Usability and Satisfaction)
  2. Device design/labeling assessments

CONTACTS AND LOCATIONS:
Overall Officials: Steven Steinhubl, MD, Principal Investigator — STSI
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States